CLINICAL TRIAL: NCT04360655
Title: A Randomized, Prospective Study of the Efficacy and Safety of the 1st Treatment in Advanced Central NSCLC by PD-1/PD-L1 Inhibitor and Chemotherapy With/Without Bronchoscopic Microwave Intervention
Brief Title: Bronchoscopic Microwave Intervention Treatment in Advanced Central NSCLC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Caicun Zhou, Director, Head of Oncology, Principal Investigator, Clinical Professor, Shanghai Pulmonary Hospital, Shanghai, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Surpass
Record Dates: First submitted 2020-04-20; First posted 2020-04-24 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Effect Increased; Safety Issues
Keywords: anti-PD-1 / PD-L1 monoclonal antibody; chemotherapy; bronchoscopic microwave intervention; advanced central non-small cell lung cancer patients
MeSH Terms: interventions — Drug Therapy; Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- anti-PD-1 / PD-L1 monoclonal antibody and chemotherapy (Active Comparator): anti-PD-1 / PD-L1 monoclonal antibody and chemotherapy
  Interventions: Drug: anti-PD-1 / PD-L1 monoclonal antibody and chemotherapy
- combined with bronchoscopic microwave intervention (Experimental): anti-PD-1 / PD-L1 monoclonal antibody and chemotherapy combined with bronchoscopic microwave intervention
  Interventions: Procedure: bronchoscopic microwave intervention; Drug: anti-PD-1 / PD-L1 monoclonal antibody and chemotherapy

INTERVENTIONS:
Procedure: bronchoscopic microwave intervention — bronchoscopic microwave intervention
  Other Names: Local treatment
  Arms: combined with bronchoscopic microwave intervention
Drug: anti-PD-1 / PD-L1 monoclonal antibody and chemotherapy — anti-PD-1 / PD-L1 monoclonal antibody and chemotherapy
  Other Names: Systemic treatment

SUMMARY:
A randomized, prospective study of the efficacy and safety of the first-line treatment in advanced central non-small cell lung cancer patients by anti-PD-1 / PD-L1 monoclonal antibody and chemotherapy versus anti-PD-1 / PD-L1 monoclonal antibody and chemotherapy combined with bronchoscopic microwave intervention

DETAILED DESCRIPTION:
This study is a randomized, prospective study, which will analyze the efficacy and safety of the first-line treatment in advanced central non-small cell lung cancer patients by anti-PD-1 / PD-L1 monoclonal antibody and chemotherapy versus anti-PD-1 / PD-L1 monoclonal antibody and chemotherapy combined with bronchoscopic microwave intervention. The efficacy will include objective response rate, disease control rate, progression-free survival, and overall survival. The safety will include adverse events and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* advanced central non-small cell lung cancer patients, untreated, tolerating bronchoscopy

Exclusion Criteria:

* contraindications to tracheoscopy, chemotherapy, and immunotherapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-05-01 (Estimated); Primary Completion 2022-04-30 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
objective response rate | 6 weeks
  objective response rate
progression-free survival | 1 years
  progression-free survival

SECONDARY OUTCOMES:
disease control rate | 6 weeks
  disease control rate
overall survival | 2 years
  overall survival
adverse events | 3 weeks
  adverse events
quality of life score | World Health Organization Quality of Life Scale-Brief (WHOQOL-BREF)score 0-100，higher scores mean a better outcome.
  quality of life score

CONTACTS AND LOCATIONS:
Overall Officials: Caicun Zhou, MD, PHD, Principal Investigator — Shanghai Pulmonary Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No